CLINICAL TRIAL: NCT02696135
Title: The Chinese Hypertrophic Cardiomyopathy Study(CHCS)
Acronym: CHCS
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lei.Song@NCCD, MD.&ph.D, China National Center for Cardiovascular Diseases
Other Study IDs: CHCS
Record Dates: First submitted 2016-01-26; First posted 2016-03-02 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: hypertrophic cardiomyopathy; clinical outcomes; multi-omics; risk stratification
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens retained include blood, serum, plasma, and myocardium when the patients receive cardio myectomy surgery.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypertrophic cardiomyopathy: Individuals with an unexplained maximal left ventricle wall thickness ≥15 mm on echocardiography and/or cardiac magnetic resonance imaging or or ≥13 mm for individuals with family history of HCM, in the absence of other cardiac or systemic diseases capable of producing that magnitude of cardiac hypertrophy.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is one of the most common inherited cardiac diseases, with a prevalence of ∼0.2%. Sudden cardiac death (SCD), heart failure and stroke are the major poor outcomes of HCM. Although about half of the patients were found to be caused by mutations mainly located in genes encoding sarcomere proteins, the causes in a significant proportion of patients with HCM are still unknown. Even in the patients with sarcomere mutations, the molecular pathways that eventually lead to cardiac hypertrophy are remained to be revealed. Furthermore, HCM presents with significant heterogeneity. SCD risk stratification and prevention by ICD are necessary. However, the strategy of SCD risk stratification recommended by the 2011 ACCF/AHA and 2014 ESC guidelines were based mainly on the evidence derived from American and European countries. The accuracy of these guidelines in Chines patients with HCM was not evaluated yet.

DETAILED DESCRIPTION:
In the present study, patients with HCM are recruited prospectively after informed consent was given. The investigator will collect the baseline clinical characteristics of the patients at enrollment, including comprehensive physical examination, laboratory testing of blood and urine, electrocardiography, 24-hr Holter, echocardiography, MRI and other examinations if necessary. The specimens retained include blood for all patients and myocardium for patients receive surgery of myocardial myectomy. Multi-omics screening, including genomics, epigenomics, transcriptomics, proteomics, metabolomics, will be performed to identified novel disease genes, signal pathway or processes, genetic risk factors and potential therapy targets of HCM. Furthermore, besides examining the accuracy of SCD risk prediction of the 2011 ACCF/AHA and 2014 ESC guidelines, we will identify novel risk factors associated with the clinical outcomes and construct predictive models suitable for Chinese patients with HCM.

ELIGIBILITY:
Inclusion criteria: Patients with HCM diagnosed by observation of unexplained maximal left ventricle wall thickness ≥15 mm on echocardiography and/or cardiac magnetic resonance imaging or or ≥13 mm for individuals with family history of HCM.

Exclusion criteria: Individuals with other cardiac or systemic diseases capable of producing that magnitude of cardiac hypertrophy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HCM are recruited from multiple centers in China between March 23, 2016 and December 31, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-03-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular deaths | an average of 2 years
  Including SCD and deaths due to heart failure and stroke.

SECONDARY OUTCOMES:
all-cause mortality | an average of 2 years.
  deaths due to all causes.
Heart failure | an average of 2 years
  Progress to level III or IV in New York Heart Association class.
Stroke | an average of 2 years
  including cerebral infarction and hemorrhage
Malignant arrhythmia | an average of 2 years
  The incidence rate of malignant arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Song Lei, MD.&ph.D, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided